CLINICAL TRIAL: NCT06551480
Title: Pilot Study on VCSEL-based Optical Swept Source Biometry
Brief Title: VCSEL Based Optical Swept Source Biometry
Acronym: VBOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rainer Leitgeb (Other)
Collaborators: Mein Hanusch-Krankenhaus (Other)
Responsible Party: Sponsor-Investigator, Rainer Leitgeb, Prof. Dr. Rainer Leitgeb, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MUW_VBOB
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Myopia
MeSH Terms: conditions — Cataract; Myopia | interventions — Biometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Study (Experimental): Pilot study in healthy participants and cataract patients
  Interventions: Device: Biometry

INTERVENTIONS:
Device: Biometry — Only one eye from each patient will be included in the study. All subjects and patients included in the study will undergo biometric measurements with both devices (IOL master 500 and VCSEL based swept source optical biometry).

SUMMARY:
Optical interferometric biometry is a non-invasive and highly precise method for measuring eye length and intraocular distances. The method already exists as commercial devices (e.g. IOLMaster, Carl Zeiss Meditec AG). A major cost factor of the devices available on the market is the laser used. The use of a much cheaper laser could significantly reduce the price of these devices, which would lead to greater availability of this technology in developing countries. This would make it possible to replace the ultrasound methods used to date and thus enable contact-free measurements, which in turn can reduce the spread of infectious diseases.The study investigates the use of a thermally tunable vertical cavity surface emitting laser (VCSEL) for optical swept source biometry.

DETAILED DESCRIPTION:
1. Background

   With 15 million operations per year, cataract surgery is the most commonly performed eye surgery. The number of operations worldwide is expected to increase by 25% between 2008 and 2015.

   The simplest operation is the implantation of a monofocal intraocular lens (IOL). It is the most commonly performed cataract procedure in developing countries (e.g. 65% in India), as well as in rural and poor areas in industrialized countries. To prepare for the operation, simple IOL calculation formulas are used that require knowledge of the axial eye length. Today, biometry is mainly performed by applanation ultrasound and simple keratometers. However, optical measurement by low coherence interferometry (OCT) is becoming increasingly important, as it has the important advantage of being contact-free and thus avoiding complications that can be caused by possible infections. In addition, the method is extremely precise and does not depend on the skill of the doctor. A major cost factor in the production of such devices is the laser used. The use of a much cheaper laser diode could significantly reduce the price, which would ensure availability even in developing countries.
2. Rationale The suitability of electrically tuned VCSEL laser diodes as light sources for determining intraocular distances is to be investigated. The results are to be compared with those of a commercial device in terms of signal quality and measurement accuracy. Such a device would be contact-free, which would help prevent infections, would be significantly cheaper than currently available methods, and would be able to determine intraocular distances very precisely.
3. Study objectives The aim of the study is to demonstrate the usability of an electrically tuned VCSEL laser diode as a cost-effective alternative to the lasers used to date. To this end, the precision, reproducibility and manageability of the measurement with the VCSEL laser diode will be investigated. Test subjects and cataract patients will be examined. The precision of the measurement with the device of intraocular distances will be compared with that of a commercial device, IOLMaster500 from Carl Zeiss Meditec.
4. Study Design

The study is a pilot study. It takes the measurement principle of a commercially available device for measuring eye length as a starting point.

The technology used is swept source Optical Coherence Tomography. This swept source is to be implemented using the electrically tuned VCSEL laser diode. Such laser diodes are able to change their central wavelength by changing the driver current. Another advantage arises from the VCSEL technology used in the laser diode used. This type of laser diode has a very narrow instantaneous line width and thus a very long coherence length, which far exceeds that required for the biometry of the eye.

In swept source OCT, the attenuation of the signal in depth is much lower than in spectrometer-based systems. In addition, the sensitivity is higher than with time-domain partial coherence interferometry (PCI) biometry systems and they are much faster. The reason is that the entire axial structure is encoded in parallel in the spectrum.

4.1. Implementation and evaluation: In the proposed study, intraocular distances, primarily the axial eye length and the anterior chamber depth, of the participating subjects and patients are to be determined using the method described. This is an exploratory pilot study to determine whether the VCSEL-based technology is suitable (in terms of speed of measurement and sensitivity of the method) to achieve a precise determination of the axial eye length in both healthy subjects and cataract patients with various degrees of cataract. The measurements with the IOLMaster serve as a basis for comparison.

Participants in the study are to be healthy subjects and cataract patients. All participants will first undergo a routine examination. Other risks will also be identified during the routine examination. These examinations will be carried out at the Eye Clinic.

The test subjects and patients are then measured using the measurement setup at the Center for Medical Physics and Biomedical Engineering.

The routine examination at the eye clinic includes a slit lamp and eye length measurement. The eye to be examined is selected by the investigator during the routine examination.

4.2 Selection of the study population The participants are recruited via public notices. 30 healthy subjects are selected between the ages of 19 and 85 years. 30 cataract patients are selected between the ages of 19 and 85 years .

4.3 Preliminary examination:

* Routine examination at the Eye Clinic of the Medical University of Vienna. - - Measurement of eye length using IOL Masters.
* For cataract patients, the degree of cataract is determined based on the Lens Opacities Classification Systems (LOCS III)

4.4. Withdrawal or replacement of study participants

The study participants will be excluded from the study under the following circumstances:

* If they so wish
* If the study director believes that the study is not in the interest of the study participant
* If the study participant violates one of the requirements and points of the consent form In any case, the study exclusion will be recorded with a detailed explanation. If the study has to be terminated, the data will be retained.

Study participants who cannot complete the study will be replaced. The data can, however, be used for analysis.

4.5. Target variables

Axial eye length and anterior chamber depth: standard deviation and mean over repeated measurements will be analyzed; A comparison with the reference device will be established through Bland-Altman analysis.

Measurements are taken per study participant with IOL Master (Carl Zeiss Meditec AG) and measurement setup with current tuned VCSEL diode

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* cataract patients (LOCS III grading)
* written informed consent

Exclusion Criteria:

* corneal pathology that would significantly influence biometric measurements
* pathologies that could affect fixation abilities other than cataract
* pregnancy (for women in reproductive age a pregnancy test will be performed)

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
axial length | 1 day
  limits of agreement between the optical biometers (mm)
anterior chamber depth | 1 day
  limits of agreement between the optical biometers (mm)

SECONDARY OUTCOMES:
intraocular distances | 1 day
  repeatability on the VCSEL swept source biometer for axial length, anterior chamber depth, corneal thickness, and lens thickness

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Leitgeb, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
All results will be shared in a published paper.